CLINICAL TRIAL: NCT05616767
Title: Prevention and Screening for Early Detection of HPV-related Cancers in Gay and Bisexual Men in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 000017185
Record Dates: First submitted 2022-10-28; First posted 2022-11-15 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: HPV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training on self-screening and HPV vaccination administration (Experimental): teaching SMM in Tanzania to conduct self-exams for oropharyngeal hrHPV-associated cancers using cellphone-mediated oral selfies, and administering the HPV vaccination series (with 2 and 6-8 month follow-up) to those who request it
  Interventions: Other: Training on self-screening and HPV vaccination administration

INTERVENTIONS:
Other: Training on self-screening and HPV vaccination administration — Participants will be taught how to do self-screening for HPV-associated cancers using Training on self-screening and HPV vaccination administration. They will also be given HPV vaccination series.

SUMMARY:
The long-term objective of the parent study is "to reduce the effects of OPCa through secondary prevention (i.e., early detection, diagnosis and treatment referral)." Consistent with this, this supplement will test HPV-related interventions tailored for Sexual Minority Men (SMM). Acceptability, feasibility and preliminary effectiveness of a smart-phone delivered Oropharyngeal Cancer (OPCA) self-assessment tool will be assessed. Given that homosexuality is stigmatized and criminalized in Tanzania, and that cell phone use is the key way SMM communicate in Tanzania, a self-assessment screening cell phone intervention holds particular promise for SMM in Tanzania but warrants separate evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* gay or bisexual men
* speak Kiswahili or English
* resident in Dar es Salam

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gay or bisexual men
Enrollment: 83 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
assess screening practices of hrHPV-related OPCa | Baseline
  Questionaire
To assess the acceptability and feasibility of teaching SMM in Tanzania to conduct self-exams | baseline to 6 months
  Questionaire to assess post-test selfie evaluations, Scores: 0= was not trained; 1= was trained; 2=took a selfie; 3= clear selfie
To assess the acceptability and feasibility of hrHPV vaccination | baseline
  percentage of individuals recruited for aim 1 who request HPV vaccination, Scores are 0=no vaccination; 1=first vaccination; 2= second vaccination; 3=third vaccination
To assess the acceptability and feasibility of hrHPV vaccination | 1 month
  percentage of individuals recruited for aim 1 who request HPV vaccination, Scores are 0=no vaccination; 1=first vaccination; 2= second vaccination; 3=third vaccination
To assess the acceptability and feasibility of hrHPV vaccination | 6 months
  percentage of individuals recruited for aim 1 who request HPV vaccination, Scores are 0=no vaccination; 1=first vaccination; 2= second vaccination; 3=third vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Dar es Salaam, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No